CLINICAL TRIAL: NCT01892410
Title: 100 Human Subject Repeat Insult Patch Test Skin Irritation/Sensitization Evaluation (Semi-Occlusive Patch)
Brief Title: Patch Test Skin Irritation/Sensitization of Cetaphil Restoraderm Skin Restoring Body Wash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04.SRE.US10235
Record Dates: First submitted 2013-06-25; First posted 2013-07-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2013-06

CONDITIONS: Skin Irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetaphil Restoraderm Skin Restoring Body Wash (Experimental): All subjects receive Cetaphil Daily Advance Ultra Hydrating Lotion
  Interventions: Other: Cetaphil Restoraderm Skin Restoring Body Wash

INTERVENTIONS:
Other: Cetaphil Restoraderm Skin Restoring Body Wash — Diluted (10%) 0.2ml or 0.2g of Cetaphil on semi-occlusive, hypoallergenic patch applied to skin for 24 hrs 9 times on Monday, Wednesday, and Friday for 3 weeks

SUMMARY:
Determine if Cetaphil Restoraderm Skin Restoring Body Wash proves to be a contact sensitizer or irritant in certain individuals.

ELIGIBILITY:
Inclusion Criteria:

* Not currently under a doctor's care
* Free of dermatological or systemic disorder which would interfere with the results
* Free of any acute or chronic disease
* Will complete a preliminary medical history form and are in general good health
* Can read, understand, and sign informed consent

Exclusion Criteria:

* Under 18 years old
* Currently under doctor's care
* Currently taking any medication
* History of acute or chronic disease
* Diagnosed with chronic skin allergies
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Area of irritation measured to determine sensitivity | 3 weeks
  9 consecutive 24hr exposures for every Monday, Wednesday, and Friday for 3 consecutive weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mayya Tastene, MD, Principal Investigator — AMA Laboratories
Locations (1):
- AMA Laboratories, Inc., New City, New York, United States